CLINICAL TRIAL: NCT00536575
Title: Phase I/II Trial of Sorafenib and Weekly Bortezomib in the Treatment of Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Sorafenib and Bortezomib Treatment for Relapsed or Refractory Multiple Myeloma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MM 14
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Results first posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed; Refractory; Sorafenib; Bortezomib
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Bortezomib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): The trial was designed as a single-arm Phase I/II study of sorafenib and bortezomib with dose optimization in initial patients. Phase I consisted of cohorts of 3 patients at each of three dose levels. Patients received bortezomib (Dose Level 1 - 1.3 mg/m2; Dose Level 2 - 1.6 mg/m2) by IV bolus on days 1, 8, 15, and 22 of each 5-week cycle with continuous oral dosing of sorafenib at 200 mg twice daily. Dose level 3 was planned as bortezomib 1.6 mg/m2 IV bolus on days 1, 8, 15, and 22 with sorafenib 400 mg by mouth twice daily throughout each 5-week cycle.
  Interventions: Drug: Bortezomib; Drug: Sorafenib

INTERVENTIONS:
Drug: Bortezomib — Dose Level 1: Bortezomib 1.3mg/m2 IV bolus on days 1, 8, 15, and 22 of each 5-week cycle.
  Dose Level 2: Bortezomib 1.6 mg/m2 IV bolus on days 1, 8, 15, and 22 of each 5-week cycle.
  Dose Level 3: Bortezomib 1.6mg/m2 IV bolus on days 1, 8, 15, and 22 of each 5-week cycle.
  Other Names: Velcade
Drug: Sorafenib — Dose Levels 1 and 2: 200 mg by mouth twice daily
  Dose Level 3: 400 mg by mouth twice daily
  Other Names: Nexavar

SUMMARY:
This is a single-arm Phase I/II study of sorafenib and bortezomib with dose optimization in initial patients. The initial patients on the dose-finding portion of this study will be enrolled through a single institution. Following establishment of the Phase II dose the study will open enrollment throughout the Sarah Cannon Research Institute (SCRI) Oncology Research Consortium.

The purpose of this study is to develop the combination of bortezomib (which is proven to be clinically active in patients with multiple myeloma) with sorafenib (a potent inhibitor of angiogenesis). This regimen will be developed in a schedule that is convenient for patients, and that is as minimally toxic to patients as possible.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the efficacy of sorafenib with weekly bortezomib, as measured by objective response rate and progression-free survival in patients with relapsed/refractory multiple myeloma.

Secondary Objective:

To evaluate the feasibility and toxicity of sorafenib with weekly bortezomib in the treatment of patients with relapsed/refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must have been previously diagnosed using standard criteria and have received no more than 2 prior regimens for the treatment of multiple myeloma.
* Participant must be defined as Relapsed or Refractory Disease by one of the following criteria prior to enrollment: Relapsed Disease after high-dose therapy (autologous stem cell transplantation) as part of the first-line line treatment program. These patients may have received a maximum of 1 previous regimen, Refractory Disease or Relapsed Disease after > 1 prior therapy for multiple myeloma. Prior bortezomib treatment permitted if the patient achieved a documented response.
* ECOG performance status 0, 1, or 2.
* WBC >= 3000; ANC >= 1000; platelets >= 50,000 (Patients with platelets >= 30,000 are eligible if thrombocytopenia is felt to be due to extensive bone marrow involvement with myeloma).
* Serum creatinine < 2.0 mg/dL for a calculated or measured creatinine clearance > 30 mL/minute
* Total bilirubin < 1.5 x ULN
* ALT and AST < 2.5 x the ULN ( < 5 x ULN for patients with liver involvement)
* INR < 1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Patients must have measurable or evaluable disease. In patients with disease limited to bone and bone marrow, serial paraprotein measurements are acceptable for evaluable disease.

Exclusion Criteria:

* Patients with > grade 1 peripheral neuropathy.
* Thrombolic or embolic events such as a cerebrovascular accident, including transient ischemic attacks, within the past 6 months.
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Known brain metastasis. Patients with neurological symptoms must undergo CT scan/MRI of the brain to exclude brain metastasis.
* Patients with other medical conditions that would potentially interfere with their participation in this trial.
* Patients with other active malignancies, or history of treatment for other invasive cancers, within 3 years of study entry.
* Patients with previous evidence of hypersensitivity to sorafenib, bortezomib, boron, or mannitol.
* Women who are pregnant or lactating are ineligible. All patients of childbearing potential are required to use adequate methods of contraception while receiving study treatment, and for at least 2 weeks after the last dose of sorafenib. Men should continue to use contraception until at least 3 months after their last dose of sorafenib.
* Evidence of POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome.
* Cardiac disease: Congestive heart failure > class II NYHA (see Appendix D.) Patients must not have unstable angina (anginal symptoms at rest), new onset angina (began within the last 3 months), or myocardial infarction within the past 6 months.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection > CTCAE Grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-11; Primary Completion 2010-02 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian W. Flinn, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (2):
- United States (2):
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- See also: Sarah Cannon Research Institute — http://www.sarahcannonresearch.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib/Bortezomib: The trial was designed as a single-arm Phase I/II study of sorafenib and bortezomib with dose optimization in initial patients. Phase I consisted of cohorts of 3 patients at each of three dose levels. Patients received bortezomib (Dose Level 1 - 1.3 mg/m2; Dose Level 2 - 1.6 mg/m2) by IV bolus on days 1, 8, 15, and 22 of each 5-week cycle with continuous oral dosing of sorafenib at 200 mg twice daily. Dose level 3 was planned as bortezomib 1.6 mg/m2 IV bolus on days 1, 8, 15, and 22 with sorafenib 400 mg by mouth twice daily throughout each 5-week cycle.
Period: Overall Study
Arm/Group | Sorafenib/Bortezomib
Started | 13
Completed | 11
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib/Bortezomib
Number analyzed (Participants) | 13
Age Continuous [Median (Full Range); unit: years] | 67 [41 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: The percentage of patients who experience an objective benefit from treatment, determined by the treating physician after reviewing key laboratory values from blood and urine.
Time Frame: 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib/Bortezomib
Number analyzed (Participants) | 11
percentage of participants | 15

ADVERSE EVENTS:
Arm/Group | Sorafenib/Bortezomib
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib/Bortezomib (N=13)
Cardiopulmonary Arrest (Cardiac disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Death (General disorders) | 1 (1)
Infection - Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sorafenib/Bortezomib (N=13)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3)
Amyloidosis (General disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (11)
Bilirubin (Metabolism and nutrition disorders) | 1 (1)
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 (1) — Bradycardia
Cardiopulmonary Arrest (Cardiac disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Cold Symptoms (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Death (General disorders) | 1 (1)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 3 (6)
Diarrhea (Gastrointestinal disorders) | 4 (11)
Disease Progression (General disorders) | 1 (2)
Dizziness (Nervous system disorders) | 2 (4)
Dry Eye (Eye disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema (Blood and lymphatic system disorders) | 3 (4)
Creatinine (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 10 (29)
Fever (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1/1 (1)
Glaucoma (Eye disorders) | 1 (1)
Hand-Foot (Skin and subcutaneous tissue disorders) | 5 (8)
Heartburn (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 9 (26)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) — Nosebleed
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Cardiac disorders) | 4 (7)
Hyperviscosity (Blood and lymphatic system disorders) | 1 (1)
Hypogammaglobulinemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Infection - Other (Infections and infestations) | 6 (8)
Insomnia (General disorders) | 2 (2)
Joint - Effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytes (Immune system disorders) | 7 (17)
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 3 (9)
Nausea (Gastrointestinal disorders) | 5 (9)
Altered mental status (Nervous system disorders) | 1 (1)
Neuropathy - Motor (Nervous system disorders) | 1 (1)
Neuropathy - Peripheral (Nervous system disorders) | 1 (1)
Neuropathy - Sensory (Nervous system disorders) | 6 (17)
Neutrophils (Immune system disorders) | 5 (11)
Ocular - Other (Eye disorders) | 2 (2)
Pain - Other (cramp) (General disorders) | 1 (1)
Pain - Headache (General disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 5 (9)
Somnolence (General disorders) | 1 (1)
Supraventricular Arrhythmia (Cardiac disorders) | 1 (1) — atrial fibrillation
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Pain - Leg (General disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 7 (22)
Urinary Frequency (Renal and urinary disorders) | 2 (4)
Urine Color Change (Renal and urinary disorders) | 1 (1)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (4)
Weakness (General disorders) | 2 (2)
Dry skin (General disorders) | 1 (1)
Pain - abdomen (General disorders) | 1 (1)
Pain - back (General disorders) | 2 (2)
Pain - bone (General disorders) | 2 (3)
Pain - breast (General disorders) | 1 (1)
Pain - chest (General disorders) | 1 (1)
Pain - ear (General disorders) | 1 (6)
Pain - Extremity-limb (General disorders) | 7 (12)
Pain - joint (General disorders) | 3 (5)
Pain - muscle (General disorders) | 1 (2)
Pain - skin (General disorders) | 1 (2)
Pain - teeth (General disorders) | 1 (1)
Pain - throat (General disorders) | 1 (1)
Pain NOS (General disorders) | 1 (1)
Paranasal sinus reaction (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pulmonary/Upper Respiratory - other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The 15% response rate was substantially lower than the designed rate of 60% for this trial. Coupled with the influx of new compounds for the treatment of multiple myeloma it was decided that this study should be closed early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.